CLINICAL TRIAL: NCT04766320
Title: A Clinical Safety and Efficacy Study on TIL for the Treatment of r/r Gynecologic Tumors
Brief Title: Study on TIL for the Treatment of r/r Gynecologic Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Shanghai Juncell Therapeutics (Industry)
Responsible Party: Principal Investigator, Zhongping Cheng, Director of Department of Gynecology and Obstetrics, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: shiyuanfuke000
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (TIL) (Experimental): 1x10^9-3x10^11 in vitro expanded autologous TILs will be infused i.v. to patients with relapsed/refractory malignant gynecological tumors after NMA lymphodepletion treatment with fludarabine and cyclophosphamide. PD-1 checkpoint inhibitor would be applied as combination treatment to those patients.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — Adoptive transfer of 1x10^9-3x10^11 autologous TILs to patients i.v. in 30-120 minutes.

SUMMARY:
This study is to investigate the safety and efficacy of tumor infiltrating lymphocyte (TIL) therapy in patients with malignant refractory/relapsed gynecologic tumors. Autologous TILs are expanded from tumor resections or biopsies and infused i.v. into the patient after NMA lymphodepletion treatment with fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years to 75 years;
2. Histologically diagnosed as primary/relapsed/metastasized malignant tumors;
3. Expected life-span more than 3 months;
4. Karnofsky≥60% or ECOG score 0-2;
5. Test subjects have failed standard treatment regimens, or there are no standard treatment regimens available.
6. Test subjects must have tumor regions eligible for biopsy or resection, or malignant body fluid where TILs can be isolated;
7. At least 1 evaluable tumor lesion;
8. Absolute count of white blood cells≥2.5×10^9/L, absolute count of neutropils≥1.5×10^9/L, platelet count≥100×10^9, hemoglobin≥90 g/L;
9. Serum creatinine clearance 50mL/min or higher; creatinine≤1.5×ULN; ALT/AST less than three times that of normal group, ALT/AST of test subjects with liver metastasis less than five times that of normal group; bilirubin≤1.5×ULN;
10. Activated partial thromboplastin time (APTT) less than or equal to 1.5xULN; international normalized ratio (INR) less than or equal to 1.5xULN;
11. Enough venous accessibility, no absolute or relative contraindications to operation or biopsy;
12. Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent, and continue within 1 year after the completion of lymphodepletion；
13. Any malignant tumor-targeting therapies, including radiotherapy, chemotherapy and biologics must cease 28 days before obtaining TILs;
14. Be able to understand and sign the informed consent document;
15. Be able to stick to follow-up visit plan and other requirements in the agreement.

Exclusion Criteria:

1. Need glucocorticoid treatment, and daily dose of Prednisone greater than 15mg (or equivalent doses of hormones);
2. Autoimmune diseases requiring immunomodulatory treatment;
3. Serum creatinine >1.5×ULN; serum glutamic-oxalacetic transaminase (SGOT) greater than 5×ULN; bilirubin >1.5×ULN;
4. Forced expiratory volume in one second (FEV1) less than 2L, diffusing capacity of the lung for carbon monoxide (DLCO) (calibrated) less than 40%;
5. Significant cardiovascular anomalies according to any of the following definition: New York Heart Association (NYHA) Grade III or IV congestive heart failure, clinically significant low blood pressure, uncontrollable symptomatic coronary artery diseases, or ejection fraction less than 35%; Severe cardiac rhythm and conduction anomaly, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrio-ventricular conductive block, etc.
6. Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
7. Severe physical or mental diseases;
8. Blood culture positive or imaging proof;
9. Having been treated within a month or being treated now with other medicines, or other biologic therapy, chemo-or radiotherapy;
10. History of allergy to chemical compound consisting of chemical and biologic substances resembling cell therapy;
11. Having received immunotherapy and developed irAE level greater than Level 3;
12. Previous anti-tumor treatment AE did not return to CTCAE5.0 version grade 1 or below (toxicity considered by the investigator as non-safety concerns like alopecia excluded);
13. Females in pregnancy or lactation;
14. Researchers considering the test subject as having a history of other severe systemic diseases, or other reasons inappropriate for the clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is biologically possible only for females regardless of self-recognition of gender identity.
Enrollment: 15 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | Up to 12 months
  Safety assessments. Incidence of Serious Adverse Events (SAEs) and Treatment-Emergent Adverse Events (TEAEs). The severity of all adverse events was graded based on Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  To evaluate the efficacy of TIL infusion in patients as determined by objective response rate (ORR), which contains complete response (CR) and partial response (PR), using the RECIST v1.1, as assessed by the Investigator. ( CT Scan at 4-6 weeks after TIL infusion, and than every 4-6 weeks for 1 year, and then every six months after that for up to 3 years)
Disease Control Rate (DCR） | Up to 36 months
  Percentage of patients that meet CR, PR and SD criteria set in this study according to RECIST 1.1
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time length between TIL infusion and confirmed subsequent disease progression according to RECIST 1.1
Overall Survival (OS) | Up to 36 months
  The length of time from the date of the start of TIL treatment that the patients are still alive
Complete Response(CR) | Up to 36 months
  Patients with complete response per RECIST 1.1 to TIL treatment
Partial Response (PR) | Up to 36 months
  Percentage of patients with partial response per RECIST 1.1 to TIL treatment
Stable Disease (SD) | Up to 36 months
  Patients with stable disease per RECIST 1.1 to TIL treatment
Progressive Disease (PD) | Up to 36 months
  Patients with progressive disease per RECIST 1.1 to TIL treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo J, Wang C, Luo N, Wu Y, Huang W, Zhu J, Shi W, Ding J, Ge Y, Liu C, Lu Z, Bast RC Jr, Ai G, Yang W, Wang R, Li C, Chen R, Liu S, Jin H, Zhao B, Cheng Z. IL-2-free tumor-infiltrating lymphocyte therapy with PD-1 blockade demonstrates potent efficacy in advanced gynecologic cancer. BMC Med. 2024 May 20;22(1):207. doi: 10.1186/s12916-024-03420-0. PMID 38769543
- [Derived] Guo J, Luo N, Ai G, Yang W, Zhu J, Li C, Chen R, Zhang C, Liu S, Jin H, Cheng Z. Eradicating tumor in a recurrent cervical cancer patient with autologous tumor-infiltrating lymphocytes and a modified lymphodepleting regimen. J Immunother Cancer. 2022 Feb;10(2):e003887. doi: 10.1136/jitc-2021-003887. PMID 35177415